CLINICAL TRIAL: NCT05824806
Title: Knee Osteoarthritis Treatment With Platelet-rich Plasma: Prospective and Randomized Clinical Trial
Brief Title: Knee Osteoarthritis Treatment With Platelet-rich Plasma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Nacional de Traumatologia e Ortopedia (Other Government)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, Eduardo Branco de Sousa, Principal investigator, Instituto Nacional de Traumatologia e Ortopedia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 60887422.4.0000.5273
Record Dates: First submitted 2023-03-24; First posted 2023-04-24 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; platelet rich plasma; hyaluronic acid; knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in blocks by simple drawing of opaque envelopes before application, in 3 experimental groups, and identified as described below:
  GROUP A: Composed of 30 patients who will receive an intra-articular injection of platelet-rich plasma (PRP A), once a week, for three consecutive weeks; GROUP B: Composed of 30 patients who will receive an intra-articular injection of platelet-rich plasma (PRP B), once a week, for three consecutive weeks; GROUP C: Composed of 30 patients who will receive an intra-articular injection of 2 mL of intra-articular hyaluronic acid (AHI), once a week, for three consecutive weeks.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients will be randomized in block by simple drawing of opaque envelopes before application, in 3 experimental groups.
  During infiltration, patients will be sitting on the stretcher in a comfortable position, with knees flexed and blindfolded (blinding as to the treatment performed).
  Patients will be evaluated by an observer independent of the one who applied the selected treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRP protocol A (Active Comparator): Composed of 30 patients who will receive an intra-articular injection of platelet-rich plasma (PRP A), once a week, for three consecutive weeks
  Interventions: Biological: PRP Protocol A
- PRP protocol B (Active Comparator): Composed of 30 patients who will receive an intra-articular injection of platelet-rich plasma (PRP B), once a week, for three consecutive weeks
  Interventions: Biological: PRP Protocol B
- Hyaluronic acid (Placebo Comparator): Composed of 30 patients who will receive an intra-articular injection of 2 mL of intra-articular hyaluronic acid (AHI), once a week, for three consecutive weeks.
  Interventions: Device: Hyaluronic acid

INTERVENTIONS:
Biological: PRP Protocol A — Platelet rich plasma protocol A
  Arms: PRP protocol A
Biological: PRP Protocol B — Platelet rich plasma protocol B
  Arms: PRP protocol B
Device: Hyaluronic acid — Hyaluronic acid
  Arms: Hyaluronic acid

SUMMARY:
Knee osteoarthritis (KOA) is a disease characterized by cartilage degeneration, synovium inflammation, bone remodeling, osteophyte formation, inflammations and loss of articular function. Interest on biological therapies has increased due to the recent update on KOA and its natural history. Viscosupplementation with hyaluronic acid aims to restore rheological properties of synovial fluid. Platelet rich plasma (PRP) is an autologous blood product which contains an elevated platelet concentration above the one found in blood. The goal of this study is to compare the clinical results of intra articular infiltration of hyaluronic and platelet rich plasma in the treatment of KOA, and to establish a protocol for PRP obtaining and prepare. Patients form the OA treating program will be selected and randomized into three groups (treatment with hyaluronic acid or onte of the two PRP protocols, PRP A and PRP B). Evaluation will include: subjective functional evaluation, clinical evaluation, radiological evaluation and radiological evaluation, which will be performed before treatment and 3 weeks, 3 months, 6 months and 1 year after treatment. Evaluation of PRP composition will be performed using ELISA/LUMINEX.

Key words: Knee, osteoarthritis, platelet rich plasma, viscosupplementation.

DETAILED DESCRIPTION:
* The goal of the study is to compare the clinical results of infiltration with hyaluronic acid and platelet-rich plasma (PRP) in the conservative treatment of mild to moderate osteoarthritis of the knee. Besides, we want to standardize two protocols for obtaining and preparing PRP for use in the treatment of mild to moderate OA of the knee.
* The sample will consist of 90 patients with osteoarthritis of the knee being treated at the outpatient clinic of the Osteoarthritis Monitoring and Treatment Program.
* Patients will be randomized in blocks by simple drawing of opaque envelopes before application, in 3 experimental groups, and identified as described below:

GROUP PRP Protocol A: Composed of 30 patients who will receive an intra-articular injection of platelet-rich plasma (PRP A), once a week, for three consecutive weeks; GROUP PRP Protocol B: Composed of 30 patients who will receive an intra-articular injection of platelet-rich plasma (PRP B), once a week, for three consecutive weeks; GROUP Hyaluronic acid: Composed of 30 patients who will receive an intra-articular injection of 2 mL of intra-articular hyaluronic acid (AHI), once a week, for three consecutive weeks.

* PRP A will be prepared according to the following technique published previously elsewhere:

  1. Collection of 50 mL of peripheral blood from the antecubital vein, in sterile vacuum collection tubes of 5 mL with 10% sodium citrate; An aliquot of collected whole blood will be used to evaluate microbiological contamination;
  2. Centrifuge the whole blood for 10 minutes at 1200 rpm, at room temperature, separating the material into two different layers (erythrocytes, in the lower layer, and plasma, in the upper layer), in a 6.5 cm radius centrifuge;
  3. Separate and centrifuge the plasma for 5 minutes at 1200 rpm, creating two new layers (upper, which will be removed, lower, containing the platelets); Care must be taken to carefully aspirate the plasma from the closed tube using a syringe and needle and transfer it to a new collection tube, carefully injecting it through the cap;
  4. Prepare the material for infiltration in the knee; after preparation, it is estimated that 5 mL of PRP will be obtained, with half of the volume used for injection and the other half for composition analysis and microbiological analysis.
* he preparation of PRP B will be carried out according to the following technique published previously elsewhere::

  a) Collection of 50 mL of peripheral blood from the antecubital vein, in sterile vacuum collection tubes of 5 mL with 10% sodium citrate; b) Centrifuge the whole blood for 15 minutes at 1500 rpm, at room temperature, separating the material into two different layers (red blood cells, in the lower layer, and plasma, in the upper layer), in a 6.5 cm radius centrifuge; e) Separate and centrifuge the plasma for 7 minutes at 3500 rpm, creating two new layers (upper, which will be removed, lower, containing the platelets); Care must be taken to carefully aspirate the plasma from the closed tube using a syringe and needle and transfer it to a new collection tube, carefully injecting it through the cap; f) Prepare the material for infiltration in the knee; after preparation, it is estimated that 5 mL of PRP will be obtained, with half of the volume used for injection and the other half for analysis of the composition.
* All infiltrations will be performed in the outpatient procedure room using aseptic technique. The technique for application will follow the steps below:

  1. Patient sitting on the stretcher in a comfortable position, with knees flexed and blindfolded (blinding as to the treatment performed);
  2. Clean the area where the application will be performed with gauze moistened with degerming Clorhexidine;
  3. Let the chlorhexidine act for one minute and then remove it with gauze moistened with 70% alcohol;
  4. Palpation of the knee for unguided infiltration through the anterolateral approach to the knee;
  5. Perform anesthetic button on the skin and subcutaneous tissue at the infiltration site with 1 mL of 2% lidocaine without vasoconstrictor;
  6. Insert the needle attached to the syringe of the product used through the chosen path;
  7. Inject the treatment according to randomization (AHI/PRP A/PRP B);
  8. Remove the needle and empty syringe from the joint;
  9. Perform 30 knee flexion-extension cycles to distribute the product over the joint;
  10. Finalize the procedure with a simple dressing.

      * The patient should not consume fatty foods or alcoholic beverages 48 hours before the procedure;
      * If joint effusion is present, it must be aspirated before infiltration;
      * The patient should be advised to return to the hospital in case of exacerbated pain, swelling or redness in the knee;
      * NSAIDs should not be used in the week following application.
* The clinical evaluation will consist of the following steps:

  1. Subjective functional assessment, based on WOMAC questionnaires, Knee Society Score (KSS) and visual analogue scale for pain, function and satisfaction analysis (before infiltration, on the day of the third infiltration, three months, six months and one year after infiltration; according to knee center follow-up protocol);
  2. Clinical assessment, consisting of (1) registration of demographic data (age, gender, weight, height, severity of osteoarthritis), (2) range of motion measurement, (3) assessment of the axis of the lower limbs (before infiltration , on the day of the third infiltration, three months, six months and one year after the infiltration; according to the knee cernter follow-up protocol); Radiographic evaluation with panoramic, anteroposterior and profile radiographs of the knees with load, aiming to detect alterations in the axis and joint space (before infiltration, 6 months and 1 year after infiltration, according to the knee center follow-up protocol).

     Patients will be evaluated by an observer independent of the one who applied the selected treatment.
* The study of PRP composition will be carried out at the Cellular Technology Center following technique published previously elsewhere:

Peripheral blood samples from groups A and B will be processed to obtain PRP, with part of this product used in the application and part used to analyze the composition of the generated product.

Soon after preparation, a part of the product will be evaluated for hematological composition: total cell count, leukocytes and platelets, and mean platelet volume. The rest of the PRP will be stored, in aliquots of about 200ul, at the Cellular Technology Center, where it will remain frozen in a freezer at -80°C until the proteomic analysis (specified below) and the quantification of the factors and cytokines, through enzime linked immunoabsorbant assay and Luminex Kits: interleukin-1β, interleukin-6, interleukin-8, tumor necrosis factor-α, interferon-γ, interleukin-2, interleukin-2R, interleukin-7, interleukin-15, interleukin-17, interleukin-12p40 (pro-inflammatory cytokines); interleukin-1RA, interleukin-4, interleukin-5, interleukin-10, interleukin-13, interferon-α (anti-inflammatory cytokines); eotaxin, Interferon-gamma inducible Protein 10kDa, Membrane cofactor protein-1, interferon-γ-induced monokine, Macrophage inflammatory protein-1α, Macrophage inflammatory protein-1β (chemokines); endothelium growth factor, b-fibroblast growth factor, G-colony stimulating factor, vascular endotelium growth factor, transforming growth factor-β1, transforming growth factor-β2, transforming growth factor-β3, platelet derived growth factor-AB, platelet derived growth factor-BB, insulin growth factor-1 (growth factors).

ELIGIBILITY:
Inclusion Criteria:

Will be included in the study:

* Patients aged between 40 and 60 years
* Patients with bilateral osteoarthritis of the knee according to the criteria of the American College of Rheumatology
* Patients classified by radiographs using the Kellgren-Lawrence classification ≤ III in both knees
* Patients showing complete knee range of motion (0 to 120°).

Exclusion Criteria:

Will be excluded from the study:

* Patients with a history of trauma, infection or previous surgery in the joint involved
* Patients with axial deviation of the lower limbs (varus greater than 10° or valgus greater than 15°)
* Patients with previous infiltration of the knee with corticosteroids in the last six months
* Patients with previous infiltration of the knee with hyaluronic acid in the last year
* Patients with inflammatory, autoimmune or rheumatic diseases
* Patients who used non sterois anti inflammatory drugs in the previous two weeks
* Patients with body mass index>35 kg/m2
* Patients using immunosuppressants or anticoagulants
* Patients with active neoplasia
* Patients with hematologic disorders
* Patients with secondary osteoarthritis
* Patients with hip osteoarthritis
* Patients with history of acute or chronic transmissible diseases
* Patients residing outside the metropolitan region of Rio de Janeiro.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Evolution of Western Ontario and McMaster Universities Arthritis Index over time | before infiltration, two weeks after first infiltration, three months, six months and one year after last infiltration
  Subjective pain and function score changes
Evolution of Knee society score over time | before infiltration, two weeks after first infiltration, three months, six months and one year after last infiltration
  Subjective function score changes
Evolution of Visual analog pain scale over time | before infiltration, two weeks after first infiltration, three months, six months and one year after last infiltration
  Subjective pain scale changes

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo B Sousa, MD, PhD, Principal Investigator — INTO
Locations (1):
- Instituto Nacional de Traumatologia e Ortopedia, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No